CLINICAL TRIAL: NCT05685589
Title: Pilot Randomized Controlled Trial of a Telehealth Mindfulness-based Intervention for Adolescents With Autism Spectrum Disorder and Their Caregivers
Brief Title: Mindfulness-Based Intervention for Teens With Autism Spectrum Disorder and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southwest Autism Research & Resource Center (Other)
Collaborators: Arizona State University (Other); Blue Cross Blue Shield of Arizona Foundation for Community and Health Advancement (Unknown)
Responsible Party: Principal Investigator, Nicole Matthews, Ph.D., Director of Research, Southwest Autism Research & Resource Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00016672
Record Dates: First submitted 2023-01-05; First posted 2023-01-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based Intervention (Experimental): The intervention will include weekly 90-minute group meetings held online through Zoom. Adolescents and parents will meet in separate groups and will learn about mindfulness-based strategies that can be used to manage and reduce stress, anxiety, and depression. They will also learn evidence-based strategies to complete daily guided mindfulness meditations using Ten Percent Happier, a commercially-available mobile app. Participants will be encouraged to meditate using the mobile app for at least 10 minutes each day during and after the 8-week intervention.
  Interventions: Behavioral: MINDful TIME
- Delayed Treatment Control (No Intervention): Participants will be instructed to engage in treatment as usual during their 8-week wait period. After their wait period, participants will be enrolled in the mindfulness-based intervention.

INTERVENTIONS:
Behavioral: MINDful TIME — The intervention will include weekly 90-minute group meetings held online through Zoom. Adolescents and parents will meet in separate groups and will learn about mindfulness-based strategies that can be used to manage and reduce stress, anxiety, and depression. They will also learn evidence-based strategies to complete daily guided mindfulness meditations using Ten Percent Happier, a commercially-available mobile app. Participants will be encouraged to meditate using the mobile app for at least 10 minutes each day during and after the 8-week intervention.
  Arms: Mindfulness-based Intervention

SUMMARY:
This project will evaluate the effectiveness of MINDful TIME, an 8-week mindfulness-based program designed to improve mental health in adolescents with autism spectrum disorder and their caregivers. MINDful TIME includes weekly psychoeducational group meetings conducted through videoconferencing and use of a commercially available mindfulness meditation app. The investigators predict that adolescents in the mindfulness intervention group will demonstrate increases in self-reported mindfulness and reductions in self- and parent-reported anxiety and depression relative to a delayed treatment control group. The investigators will also explore whether caregivers in the treatment group demonstrate improvements in quality of life.

DETAILED DESCRIPTION:
Interested individuals and their parent/caregiver who meet preliminary eligibility criteria during the phone screen will be scheduled for a 1-2 hour virtual study visit to complete an intake interview for study and a brief IQ test. If individuals have completed this assessment at SARRC within the last five years, they will not be re-assessed; however, they will complete a 30-minute virtual intake visit to complete the intake interview, learn about the intervention and determine if they would like to participate.

Participants in the treatment group will complete three virtual study visits (Baseline, intervention exit, 2-month follow-up), whereas participants in the delayed treatment control group will complete four virtual study visits (Baseline, wait for the period exit, intervention exit, 2 month-follow-up). After completing their second-time point (i.e., wait period exit) participants in the delayed treatment control group will be enrolled in the 8-week intervention.

The investigators anticipate that the duration of an individual participant's participation in the study from baseline data collection to study completion will be approximately 6 months. Participants may be enrolled up to 8 months prior to their baseline data collection depending on when they are recruited into the study and whether they participate in cohort 1 or cohort 2.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents must be ages 13 to 18 years
* Formal clinical or educational ASD diagnosis confirmed by the study team (i.e., review of the formal diagnostic or educational report)
* Must be willing to be randomized to a treatment or delayed treatment control group
* Must be able to attend at least 7 of the 8 group meetings
* English speaking: Adolescents and their parent/caregivers must be English-speaking because the screening and behavioral measures are in English, as well as the intervention content
* Participants must live in the state of Arizona, USA

Exclusion Criteria:

* Non-verbal participants will be excluded to ensure test compliance and increase sample homogeneity.
* Participants with IQ scores <70 will be excluded because the intervention was developed for individuals without intellectual disabilities.
* Participants with a physical disability or co-occurring condition that may prevent participation in the weekly group meetings (e.g., selective mutism; aggressive behavior; inability to participate in a 90-minute video conference meeting each week)
* Participants who report active suicidal ideation

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline in Children's Depression Inventory (CDI) Scores | Post-intervention (8 weeks); 2-month follow-up
  Parent-report measure of adolescent depressive symptoms. Scores range from 30 to 90 with higher scores indicating higher levels of depression symptoms.
Mean Change from Baseline in Multidimensional Anxiety Scale for Children (MASC) Scores | Post-intervention (8 weeks); 2-month follow-up
  Parent-report measure of adolescent anxiety symptoms. Scores range from 30 to 90 with higher scores indicating higher levels of anxiety symptoms.
Mean Change from Baseline in Child and Adolescent Mindfulness Measure (CAMM) Scores | Post-intervention (8 weeks); 2-month follow-up
  Adolescent-report measure of mindfulness. Scores range from 0 to 40 with higher scores indicating higher levels of mindfulness.

SECONDARY OUTCOMES:
Mean Change from Baseline in Beck Youth Inventories (BYI) Scores | Post-intervention (8 weeks); 2-month follow-up
  Adolescent-report measure of depression. Scores range from 0 to 90, with higher scores indicating higher levels of depression.
Mean Change from Baseline in World Health Organization-Five Wellbeing Index (WHO-5) Scores | Post-intervention (8 weeks); 2-month follow-up
  Adolescent-report measure on current well-being. Scores range from 0 to 100, with higher scores indicating better quality of life.
Mean Change from Baseline in Adaptive Behavior Assessment System (ABAS-3) Scores | Post-intervention (8 weeks); 2-month follow-up
  Parent-report measure of adolescent adaptive skills across the lifespan. Scores range from 40 to 120, with higher scores indicating better adaptive skills.
Mean Change from Baseline in Social Responsiveness Scale (SRS-2) Scores | Post-intervention (8 weeks); 2-month follow-up
  Parent-report measure of adolescent presence and severity of social impairment within autism spectrum.
Mean Change from Baseline in Behavior Rating Inventory of Executive Function (BRIEF) Scores | Post-intervention (8 weeks); 2-month follow-up
  Parent-report measure of adolescent executive function and self-regulation. Scores range from 30 to 90, with higher scores indicating higher levels of executive dysfunction.
Mean Change from Baseline in Five Facets Mindfulness Questionnaire (FFMQ) Scores | Post-intervention (8 weeks); 2-month follow-up
  Adolescent-report measure of mindfulness on observation, description, aware actions, non-judgmental inner experience, and non-reactivity. Factor scores range from 1 to 5, with higher scores indicating higher levels of mindfulness.
Mean Change from Baseline in Family Quality of Life Scale (FQOL) Scores | Post-intervention (8 weeks); 2-month follow-up
  Parent-report measure of family quality of life in family interaction, parenting, emotional well-being, physical/material well-being, and disability-related support. Scores range from 1 to 5, with higher scores indicating higher satisfaction with family quality of life.
Mean Change from Baseline in Stress Index for Parents of Adolescents (SIPA) Scores | Post-intervention (8 weeks); 2-month follow-up
  Parent-report measure of the relationship of parenting stress to adolescent characteristics, parent characteristics, the quality of the adolescent-parent interactions, and stressful life circumstances. Percentile scores range from 0 to 99, with higher scores indicating higher levels of parenting stress.

CONTACTS AND LOCATIONS:
Overall Officials: Blair Braden, Ph.D, Principal Investigator — Arizona State University; Nicole Matthews, Ph.D, Principal Investigator — Southwest Autism Research and Resource Center
Locations (1):
- Southwest Autism Research and Resource Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underlie results in a publication will be available upon request to approved researchers.
Supporting Information: Study Protocol
Time Frame: Data will be available upon request starting 6 months after publication and will remain available for 2 years.
Access Criteria: Data requests should be submitted to Dr. Nicole Matthews at nmatthews@autismcenter.org and must include study aims and purpose and a detailed analysis plan describing how the data will be used. Requests will be reviewed by Dr. Matthews and access to the data will be made available through a secure link to download the requested data.

REFERENCES:
- [Derived] Matthews NL, Mitchell MM, Honda H, Malligo A, Boyd S, Pagni BA, Blair Braden B. Pilot randomized controlled trial of MINDful TIME, a novel telehealth mindfulness-based intervention for autistic adolescents and their caregivers. Autism. 2025 Jul;29(7):1864-1882. doi: 10.1177/13623613251328484. Epub 2025 Mar 31. PMID 40160168